CLINICAL TRIAL: NCT03869502
Title: European CML Blast Crisis Register
Acronym: BlastCrisis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Annamaria Brioli, Principal Investigator, University of Jena
Other Study IDs: BlastCrisis
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chronic Myeloid Leukemia in Myeloid Blast Crisis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicentric prospective and retrospective register collecting patient with CML blast crisis diagnosed in Germany and Europe

DETAILED DESCRIPTION:
Since the advent of treatment with tyrosine kinase inhibitors (TKI), the incidence of blast crises has significantly decreased. Nevertheless, about 5% of patients diagnosed with chronic myeloid leukemia (CML) will evolve into a blast phase at some point during the course of their disease. Furthermore, despite the advances made in CML treatment, outcome of patients with blast crises are still dismal. Due to the rarity of this condition clinical trials are challenging, and collaboration between researchers both at national and international level is needed to collect a meaningful number of data.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of BCR-ABL positive CML blast crisis according to the WHO criteria:

  * Blasts 20% or more of peripheral blood white cells or bone marrow cells or
  * Extramedullary blast proliferation or
  * Large foci or clusters of blasts in bone marrow biopsy

Exclusion Criteria:

* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CML Blast crisis, either newly diagnosed or as evolution of a CML in chronic phase
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | through study completion in 2024
  how many patients survive after a blast crisis event

SECONDARY OUTCOMES:
Rate of hematologic response to treatment | through study completion in 2024
  how many patients have a hematologic response to the local standard Treatment after a blast crisis event
Rate of molecular response to treatment | through study completion in 2024
  how many patients have a molecular response to the local standard Treatment after a blast crisis event
Rate of blast crises in Europe in the era of TKI treatment | through study completion in 2024
  how many patients have blast crisis events compared to all treated CML-patients in the trial centers

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Brioli, PhD MD, Principal Investigator — Univerity of Jena
Locations (9):
- Masaryk University Hospital Brno, Brno, Czechia
- Germany (6):
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - University Hospital Jena, Jena
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Universitätsmedizin Mannheim, Mannheim
  - Universitaetsklinikum Muenster, Münster
- I. P. Pavlov First St. Petersburg State Medical University, Saint Petersburg, Russia
- National Research Center for Radiation Medicine, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: No
A joint publication is planned. But no data of trial Centers will be shared with the other trial centers.